CLINICAL TRIAL: NCT01246180
Title: Study of the Cutaneous Microcirculation: ASIC Involvement.
Brief Title: Microcirculation & ASICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr Jean Louis SAUMET, Pôle d'activité médicale-Centre Hospitalier Lyon Sud-Hospices Civils de Lyon & Laboratoire de Physiologie - FRE CNRS 3075-Université Claude Bernard Lyon 1
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2009.554
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2011-07

CONDITIONS: Physiological Conditions
Keywords: Skin, microcirculation; ASIC, pressure ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — Diclofenac; Amiloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diclofenac — diclofenac 5% vs placebo (topical application) cutaneous blood flow measurement using laser Doppler
Drug: Amiloride — amiloride 1mM vs placebo (intradermal injection) cutaneous blood flow measurement using laser Doppler

SUMMARY:
Pressure ulcers are a common and costly problem. Advancing the understanding regarding the basic pathophysiological mechanisms mediating the development of pressure ulcers will allow for better delineation of populations at risk.

Healthy skin is protected from pressure-induced ischemic damage because of the presence of pressure-induced vasodilation (PIV). In contrast, in absence of PIV, such as in diabetic patients or older subjects with sensory neuropathy, the skin is exposed to severe cutaneous ischemia, which could lead to pressure ulcer formation.

Since Acid Sensing Ion channels (ASICs) appear to be involved in the cutaneous mechanosensitivity, the investigators hypothesized that PIV could be altered by treatments that block ASICs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females aged between 18 and 40 years of age

Exclusion Criteria:

* no consent, diabetes, neuropathy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
evaluate the difference in the cutaneous microvascular response to local pressure application between treated (amiloride and diclofenac) and untreated skin. | Criteria will be measured 30 and 60 minutes following the injection of amiloride and the application of diclofenac, respectively.

SECONDARY OUTCOMES:
Evaluate difference in the cutaneous sensitivity and the cutaneous microvascular response to acetylcholine, sodium nitroprusside, electrical current and local heating between treated (amiloride and diclofenac) and untreated skin | Criteria will be measured 30 and 60 minutes following the injection of amiloride and the application of diclofenac, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Saumet, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Pôle d'activité medicale-Centre Hospitalier Lyon Sud-Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Result] Fromy B, Lingueglia E, Sigaudo-Roussel D, Saumet JL, Lazdunski M. Asic3 is a neuronal mechanosensor for pressure-induced vasodilation that protects against pressure ulcers. Nat Med. 2012 Aug;18(8):1205-7. doi: 10.1038/nm.2844. Epub 2012 Jul 29. PMID 22842475